CLINICAL TRIAL: NCT00805337
Title: Compassionate Treatment of Advanced Cancer With Amplitude-Modulated Electromagnetic Fields
Brief Title: Low Levels of Electromagnetic Fields to Treat Advanced Cancer
Acronym: ADLG3
Status: No longer available | Type: Expanded Access
Sponsor: Pasche, Boris, M.D. (Individual)
Responsible Party: Boris Pasche, Cabinet Avenue de la gare 6, CH-1003-Lausanne
Other Study IDs: ADLG3
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Cancer
Keywords: Cancer amplitude-modulated electromagnetic fields
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Device: Intrabuccally-administered amplitude-modulated RFEM — Generation of amplitude-modulated electromagnetic fields: the device consists of a battery-driven radiofrequency (RF) electromagnetic field generator connected to a 1.5 meter long 50 Ohm coaxial cable, to the other end of which a spoon-shaped mouthpiece made of steel is connected with the inner conductor. The RF source of the device corresponds to a high-level amplitude-modulated class C amplifier operating at 27.12 MHz. The modulation frequency can be varied between 0.01 Hz and 150 kHz with a modulation depth of 85 ± 5%. The RF output is adjusted to 100 mW into a 50 Ohm load using a sinusoidal modulated test signal, which results in an emitting power identical to that of the device used in the treatment of insomnia (Pasche et al 1996, 19:327-336).
  Other Names: Symtonic TheraBionic

SUMMARY:
Following the discovery of tumor-specific frequencies in patients with advanced cancer, compassionate treatment with tumor-specific frequencies administered at levels that are significantly below the levels generated by cell phone will be offered to patients with limited therapeutic options.

DETAILED DESCRIPTION:
We have previously shown that the intrabuccal administration of low and safe levels of electromagnetic fields, amplitude-modulated at a frequency of 42.7 Hz by means of a battery-powered portable device modifies the electroencephalographic activity of healthy subjects (1, 2) and is associated with subjective and objective relaxation effects (3). These results prompted us to study the effects of the 42.7 Hz frequency in patients suffering from insomnia. A randomized control trial did not reveal any difference between 42.7 Hz treatment and placebo (4) but sequential administration of four insomnia-specific frequencies, including 42.7 Hz, resulted in a significant decrease in sleep latency and a significant increase in total sleep time in patients suffering from chronic insomnia (5). Dosimetric studies have shown that the amount of electromagnetic fields delivered to the brain of patients with this approach is 100 to 1000 times lower than the amount of electromagnetic fields delivered by handheld cellular phones and do not result in any heating effect within the brain (4). The U.S. FDA has determined that such a device is not a significant risk device. Lastly, a long-term follow-up survey of 807 patients who have received this therapy revealed that the rate of adverse reactions were low and were not associated with increases in the incidence of malignancy or coronary heart disease (6).

Given the advantageous safety profile of athermal, non-ionizing radiofrequency electromagnetic fields and the emerging evidence that low levels of electromagnetic or electric fields may modify the growth of tumor cells (7-9), we decided to test the hypothesis that low levels of electromagnetic fields modulated at tumor-specific frequencies may alter the growth of human malignancies. We have developed a novel patient-based biofeedback method with the goal to identify cancer-specific frequencies and have examined patients with this approach. Following identification of such frequencies in a total of 163 patients, we will offer compassionate treatment to 28 patients with advanced cancer and limited palliative therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with advanced disease and limited therapeutic options

Exclusion Criteria:

* Any patient with curative treatment options

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Kelly TL, Kripke DF, Hayduk R, Ryman D, Pasche B, Barbault A. Bright light and LEET effects on circadian rhythms, sleep and cognitive performance. Stress Med. 1997 Oct;13(4):251-8. doi: 10.1002/(SICI)1099-1700(199710)13:43.0.CO;2-0. PMID 11542396
- [Background] Pasche B, Erman M, Hayduk R, Mitler MM, Reite M, Higgs L, Kuster N, Rossel C, Dafni U, Amato D, Barbault A, Lebet JP. Effects of low energy emission therapy in chronic psychophysiological insomnia. Sleep. 1996 May;19(4):327-36. doi: 10.1093/sleep/19.4.327. PMID 8776791
- [Background] Lebet JP, Barbault A, Rossel C, Tomic Z, Reite M, Higgs L, Dafni U, Amato D, Pasche B. Electroencephalographic changes following low energy emission therapy. Ann Biomed Eng. 1996 May-Jun;24(3):424-9. doi: 10.1007/BF02660891. PMID 8734063
- [Background] Reite M, Higgs L, Lebet JP, Barbault A, Rossel C, Kuster N, Dafni U, Amato D, Pasche B. Sleep inducing effect of low energy emission therapy. Bioelectromagnetics. 1994;15(1):67-75. doi: 10.1002/bem.2250150110. PMID 8155071
- [Background] Amato D, Pasche B. An evaluation of the safety of low energy emission therapy. Compr Ther. 1993;19(5):242-7. No abstract available. PMID 8275672
- [Derived] Barbault A, Costa FP, Bottger B, Munden RF, Bomholt F, Kuster N, Pasche B. Amplitude-modulated electromagnetic fields for the treatment of cancer: discovery of tumor-specific frequencies and assessment of a novel therapeutic approach. J Exp Clin Cancer Res. 2009 Apr 14;28(1):51. doi: 10.1186/1756-9966-28-51. PMID 19366446